CLINICAL TRIAL: NCT02572427
Title: Video Laryngoscopy for Enhancing and Maintaining Intubation Skills
Brief Title: Resident Training Enhanced by New Innovations: Teleintubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202043
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2016-07

CONDITIONS: Asphyxia Neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education for intubation skills (Experimental): Interventions: Training for Pediatric Advanced Life Support (PALS) and Neonatal Resuscitation Program (NRP); 7 minute excerpt from the NRP training video regarding intubation; cognitive instruction which consisted of equipment needed for intubation; hands on instruction using the Storz video laryngoscope with manikins in simulation lab.
  Interventions: Other: Education for intubation skills
- No added education for intubation skills (Active Comparator): Interventions: Training for Routine Pediatric Advanced Life Support (PALS) and Neonatal Resuscitation Program (NRP) training; no additional training for intubating newborns.
  Interventions: Other: No added education for intubation skills

INTERVENTIONS:
Other: Education for intubation skills — Routine training in neonatal resuscitation, intensive cognitive and hands on training for intubating neonates using manikins in a simulation lab.
  Arms: Education for intubation skills
Other: No added education for intubation skills — Routine training in neonatal resuscitation but no added experience in simulation lab.
  Arms: No added education for intubation skills

SUMMARY:
The overall goal of this study was to create a simulation environment with repeated practice for residents and intense, immediate feedback. Repeated simulations for neonatal resuscitation when coupled with clinical experience have been shown to improve resident confidence.The investigators sought to determine if resident exposure to individual training and video laryngoscopy using the C-MAC video laryngoscope would improve cognitive skills and decrease intubation times in a neonatal manikin. The primary outcome was time to intubation after one year. The secondary outcome was the ability to retain cognitive instruction related to intubation

DETAILED DESCRIPTION:
Objective: Tracheal intubation of infants and children is a critical lifesaving skill, but many upper level pediatric residents are unable to successfully intubate neonates or pediatric patients in a timely manner. Simulation has been shown to be effective in teaching procedural skills, but it is not known if improvements in intubation skills can persist. The investigators sought to determine if video laryngoscopy could be used to enhance resident intubation skills that would be retained for one year.

Methods: There were 67 Pediatric and Internal Medicine/Pediatric residents, levels 1-4, who completed the study and were randomized by month of service into non-intervention (NI, n= 36) and intervention (IN, n=31) groups. IN residents observed the intubation portion of the Neonatal Resuscitation Program (NRP) training video and received cognitive instruction and 30 minutes of hands on instruction using a video laryngoscope. At the study's conclusion, 12 months after enrollment, residents completed a survey of intubations of live patients over the past year, a cognitive assessment of intubation, and were timed on intubating a manikin. Results were analyzed by Student's T-Test.

ELIGIBILITY:
Inclusion criteria:

* Pediatric residents

Exclusion criteria:

* Residents from other departments
* Neonatology fellows
* Medical students
* Medical school Faculty

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Hall, M.D., Principal Investigator — University of Arkansas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education for Intubation Skills | No Added Education for Intubation Skills
Started | 37 | 45
Completed | 31 | 36
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education for Intubation Skills | No Added Education for Intubation Skills | Total
Number analyzed (Participants) | 37 | 45 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 45 | 82
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 35 | 56
  Male | 16 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 37 | 41 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 31 | 38 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 45 | 82

OUTCOME MEASURES:

1. Primary Outcome: Skill in Intubating Neonatal Manikin
Description: Time in seconds needed to intubate neonatal manikin Skill test on neonatal resuscitation in simulation lab
Time Frame: Up to two minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Education for Intubation Skills | No Added Education for Intubation Skills
Number analyzed (Participants) | 31 | 36
seconds | 23.4 (22.4) | 39.9 (38.2)
Statistical Analysis 1: Comparison: Education for Intubation Skills vs No Added Education for Intubation Skills; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

2. Secondary Outcome: Knowledge Concerning Intubation of Neonates
Description: Score on cognitive test on intubation of neonates.Scores ranged on scale from 0 to 21 , with higher score indicating greater knowledge (better outcome).
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Education for Intubation Skills | No Added Education for Intubation Skills
Number analyzed (Participants) | 31 | 36
scores on a scale | 15 (1.7) | 13.1 (2.3)
Statistical Analysis 1: Comparison: Education for Intubation Skills vs No Added Education for Intubation Skills; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Education for Intubation Skills | No Added Education for Intubation Skills
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/45
Other Adverse Events (participants affected / at risk) | 0/37 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes